CLINICAL TRIAL: NCT03609827
Title: Population Pharmacokinetics (PK) of Melphalan in Pediatric Patients Undergoing Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Study of Melphalan Drug Exposure in Pediatric Hematopoietic Stem Cell Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: P1517152; 150811 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-01-05; First posted 2018-08-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hematologic Malignancies; Nonmalignant Diseases; Immunodeficiencies; Hemoglobinopathies; Genetic Inborn Errors of Metabolism; Fanconi's Anemia; Thalassemia; Sickle Cell Disease
Keywords: Melphalan; Pharmacokinetics; Pediatric; Allogeneic
MeSH Terms: conditions — Hematologic Neoplasms; Immunologic Deficiency Syndromes; Hemoglobinopathies; Fanconi Anemia; Thalassemia; Anemia, Sickle Cell | interventions — Melphalan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing Hematopoietic Stem Cell Transplant: Children undergoing allogeneic hematopoietic stem cell transplant (alloHCT) at University of California, San Francisco Benioff Children's Hospital.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan
  Other Names: Evomela

SUMMARY:
Melphalan is a chemotherapy drug used extensively in bone marrow transplantation. The goal of this study is to determine what causes some children to have different drug concentrations of melphalan in their bodies and if drug levels are related to whether or not a child experiences severe side-effects during their bone marrow transplant. The hypothesis is that certain clinical and individual factors cause changes in melphalan drug levels in pediatric bone marrow transplant patients and that high levels may cause severe side-effects.

DETAILED DESCRIPTION:
Melphalan is an alkylating agent with potent antitumor and immunosuppressive properties used in conditioning regimens of pediatric allogeneic hematopoietic cell transplantation (alloHCT) to promote stem cell engraftment.

This is a single-center, prospective, non-interventional pharmacokinetics (PK) study investigating the clinical pharmacology of melphalan in 24 children undergoing allogeneic hematopoietic stem cell transplant (alloHCT) at University of California, San Francisco Benioff Children's Hospital.

Patients would receive melphalan regardless of whether or not they decide to consent to PK sampling.

Melphalan doses will not be adjusted based on PK data.

The investigators will apply the combination of a limited sampling strategy and population PK methodologies to determine specific factors influencing melphalan exposure in pediatric alloHCT recipients. Population PK methodologies support the use of sparse sampling and therefore allow us to investigate drug levels in a pediatric population that would otherwise not be feasible using traditional intensive PK sampling.

Subjects will undergo PK sampling of plasma melphalan drug concentrations over the duration of melphalan therapy (3 to 5 days).

To evaluate sources of variability impacting melphalan exposure clinical data will be obtained from the patient's medical chart on each day of PK sampling.

To assess exposure-response relationships neutrophil engraftment, treatment-related toxicity, and survival data will be collected through day 100 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-17 years of age
* Undergoing alloHCT for the treatment of malignant or nonmalignant disorder
* Receiving melphalan-based preparative regimen

Exclusion Criteria:

* Any child 7-17 years of age unwilling to provide assent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population for the proposed study includes children 0-17 years of age undergoing alloHCT for the treatment of malignant and nonmalignant disorders. Patients receiving melphalan over 3 to 5 days are eligible to participate. All patients enrolled in this study will undergo PK sampling on the inpatient pediatric BMT unit at UCSF Benioff Children's Hospital. The proposed research will not study any patients receiving melphalan in a clinic or any other out-patient setting.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of melphalan for HCT in pediatric patients. | 5min post end of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of melphalan for HCT in pediatric patients. | 15 min post end of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of melphalan for HCT in pediatric patients. | 30 min post end of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of melphalan for HCT in pediatric patients. | 1 hr post end of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of melphalan for HCT in pediatric patients. | 2 hrs post end of infusion

SECONDARY OUTCOMES:
Evaluate the event free survival according to the AUC of melphalan | 1month post transplant
Evaluate the event free survival according to the AUC of melphalan | 3 months post transplant
Evaluate the event free survival according to the AUC of melphalan | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Janel R Long-Boyle, PharmD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No